CLINICAL TRIAL: NCT06769438
Title: Effectiveness of the Augmented Rehabilitation of Digestive Surgical Emergencies Pathway in Reducing Unscheduled Hospitalizations After Surgery
Brief Title: Effectiveness of the RAUC Pathway in Reducing Unscheduled Hospitalizations After Emergency Digestive Surgery
Acronym: RAUCAMIENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2024_843_0094
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Digestive Emergency; New Pathway; Connected Health
Keywords: digestive emergency; new pathway; connected health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): patients included in the CHUAP RAUC + course
  Interventions: Other: ERAS; Other: ROFIM; Other: DEEPSEN; Other: RDS; Other: Get ready; Other: Lumiradx; Other: Digital Surgery
- Control group 1 (Active Comparator): patients from CHU Rouen included over the same period as patients from CHUAP benefiting from standard care (RAUC -)
  Interventions: Other: ERAS
- Control group 2 (Active Comparator): patients verifying the inclusion/non-inclusion criteria and from the SNDS over the period from January 1, 2022 to December 31, 2025
  Interventions: Other: ERAS

INTERVENTIONS:
Other: ERAS — ERAS
Other: ROFIM — teleexpertise solution connecting extra-hospital and intra-hospital practitioners
  Arms: Experimental group
Other: DEEPSEN — virtual reality headset to reduce anxiety
  Arms: Experimental group
Other: RDS — patch to continuously monitor patients' physiological parameters at home
  Arms: Experimental group
Other: Get ready — digital solution for managing patients at home
  Arms: Experimental group
Other: Lumiradx — taking CRP at home
  Arms: Experimental group
Other: Digital Surgery — recording of the different operating times
  Arms: Experimental group

SUMMARY:
The number of emergencies's visits (22 million visits in 2019 in France), the organization of emergencies and the sustainability of the current health system are threatened. In the CHUAP adult emergency department, 60,000 visits were recorded in 2022.

Unlike medical emergencies which have structured their care and research activities (heart, brain), and whose organization has demonstrated its general interest for society, digestive surgical emergencies, which involve complex patients (elderly people, comorbidities) , emergency situations and surgical procedures, have never been thought of globally in terms of personalized care and research pathways. Currently, patients treated in emergency are managed without a pre-established optimization program and without a dedicated pathway, where emergency constitutes a major risk factor for postoperative complications.

RAUCAMIENS evaluates a new care pathway implemented within the framework of the RHU RAUC : the implementation of the Enhanced rehabilitation after surgery (ERAS) and e-health devices for home monitoring, for patients treated in the emergency room for a digestive pathology. The purpose is to evaluate the effectiveness of the RAUC pathway in reducing the rate of unplanned hospitalization readmission after emergency digestive surgery 30 days postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Criterion linked to the protocol :

  -- Patient consulted in emergency for a digestive pathology requiring surgery
* Search criteria:

  * Adult patient (≥ 18 years old),
  * Able to give consent,
  * Affiliation to a social security scheme

Exclusion Criteria:

* Criterion linked to the protocol:

  * Patient leaving hospitalization to a convalescent center
  * Patient requiring direct operating room (vital emergency or surgical revision)
  * Patient presenting to the emergency room for a postoperative complication
  * Patient directly admitted to intensive care
* Search criteria:

  * Pregnant or breastfeeding woman
  * Patient under guardianship, curatorship or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Occurrence of an unscheduled hospitalization readmission | 30 days
  Occurrence of an unscheduled hospitalization readmission following digestive surgery performed urgently within 30 days

SECONDARY OUTCOMES:
Clavien-Dindo score | 30 days
Duration of hospitalization linked to the first admission to perform emergency digestive surgery | 30 days
  Duration of hospitalization linked to the first admission to perform emergency digestive surgery
Quality of life score | 0 day
  Quality of life assessed by the scores of the different dimensions of the EQ-5D-5L which is a PROMS, at admission
Quality of Life score | 30 days
  Quality of life assessed by the scores of the different dimensions of the EQ-5D-5L which is a PROMS
STAI-Y scale | 0 day
  Anxiety assessed by the STAI-Y scale
Transition to emergency without hospitalization | 30 days
  Transition to emergency without hospitalization
incremental cost-utility ratio | 30 days
  incremental cost-utility ratio
incremental cost-effectiveness ratio | 30 days
  incremental cost-effectiveness ratio (cost per readmission avoided)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc Regimbeau, Pr, Principal Investigator — CHRU Amiens
Locations (2):
- France (2):
  - CHU Rouen, Rouen
  - Centre Hospitalier Universitaire, Amiens, Salouël

IPD SHARING:
Plan to Share IPD: No